CLINICAL TRIAL: NCT04677400
Title: More Than Body Appearance (MBA) Intervention: Investigation of the Efficacy of a Psychological Online Intervention to Improve Body Image
Brief Title: More Than Body Appearance (MBA) Intervention
Acronym: MBA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Silvia Cerea, Ph.D., University of Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 3811
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-09

CONDITIONS: Body Image
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants in the Experimental group start the MBA intervention immediately (Time 0; T0).
  Interventions: Other: More than Body Appearance (MBA) Intervention
- Waiting-list group (Active Comparator): Participants in the waiting-list group start the MBA intervention at Time 1 (T1; 15 days after the Experimental group).
  Interventions: Other: More than Body Appearance (MBA) Intervention

INTERVENTIONS:
Other: More than Body Appearance (MBA) Intervention — The MBA is an online psychological intervention designed to improve body image. The intervention lasts 15 days, and it comprises two types of activity (1st and 2nd week).
  During the first week of the MBA intervention, participants sill read three blocks of psychoeducational material including information about: 1) body image; 2) positive body image and healthy lifestyles; and 3) body functionality.
  During the second week participants produce 3 structured writing assessment pertaining to body functionality and why it is important. Each assignment focused on two areas of body functionality: 1) body's senses and physical capacities; 2) health and creative skills; 3) self-care/daily routine and communication with others. For each writing assignment, participants were asked to reflect, describe, and specify why these aspects of body functionality were personally important and meaningful to them.

SUMMARY:
The promotion of a positive body image is crucial to increase the efficacy of psychological interventions targeting body image. Recent studies indicated that positive body image also acts as a protective factor against the onset of ED symptoms. However, in the last decades, research has predominantly focused on reducing body dissatisfaction, with most available psychological interventions for body image adopting a disease reduction perspective while neglecting positive aspects of psychological functioning. This approach has shown limited efficacy in improving body image. Consequently, it is crucial to develop new psychological interventions including both perspectives (i.e., disease reduction and health promotion perspectives) to improve body image and to test their efficacy in different contexts and populations.

The aim of this study was to investigate the efficacy of a 2-week online psychological intervention (More than Body Appearance; MBA) designed to improve body image in young women at both high and low risk of developing Body Image Disorders and in female athletes practicing aesthetic sports.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above

Exclusion Criteria:

* Presence of a full-blown Body Image Disorder (BID);
* Current treatment for a BID.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Body appreciation | 2 weeks
  Improvements in body appreciation assessed by means of a self-report questionnaire: Body Appreciation Scale-2 (BAS-2; Minimum value: 10; Maximum value: 50; higher scores represent higher body appreciation)
Body dysmorphic disorder symptoms | 2 weeks
  Reductions in body dysmorphic disorder symptoms assessed by means of a self-report questionnaire: Questionario sul Dismorfismo Corporeo (QDC; Minimum value: 40; Maximum value: 280; higher scores represent higher body dysmorphic disorder symptoms)
Functionality appreciation | 2 weeks
  Improvements in functionality appreciation assessed by means of a self-report questionnaire: Functional Appreciation Scale (FAS; Minimum value: 7; Maximum value: 35; higher scores represent higher body functionality)

SECONDARY OUTCOMES:
Risk of developing eating disorders | 2 weeks
  Reductions of the risk of developing eating disorders assessed by means of a self-report questionnaire: Eating Disorder Inventory-3 (EDI-3; Minimum value: 25; Maximum value: 150; higher scores represent higher risk)
Intuitive eating | 2 weeks
  Improvements in intuitive eating assessed by means of a self-report questionnaire: Intuitive Eating Sale-2 (IES-2; Minimum value: 23; Maximum value: 115; higher scores represent higher intuitive eating practices)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Cerea, PhD, Principal Investigator — Department of General Psychology, University of Padova
Locations (1):
- University of Padua, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No